CLINICAL TRIAL: NCT03421561
Title: ProspectIve, Randomized, SingLe-Blind, U.S. MuLti-Center Study to EvalUate TreatMent of Obstructive SupErficial Femoral Artery or Popliteal LesioNs With A Novel PacliTaxel-CoatEd Percutaneous Angioplasty Balloon Pivotal Post-Approval Study
Brief Title: ILLUMENATE Pivotal Post-Approval Study (PAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D035940
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DCB Subjects (Experimental): The Stellarex DCB is a commercially available PTA balloon catheter (EverCross™ 0.035" PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA) coated with paclitaxel using a proprietary carrier.
  Basic Catheter Specifications
  * Guidewire: 0.035"
  * Balloon Length: 40/80/120 mm
  * Sheath Compatibility: greater than or equal to 6 French
  * Balloon Diameter: 4/5/6 mm
  * Shaft length: 135 cm The nominal dose density of paclitaxel on the Stellarex DCB is 2.0 μg/mm2. Indications The Stellarex 0.035" OTW Drug-coated Angioplasty Balloon is indicated for percutaneous transluminal angioplasty (PTA), after appropriate vessel preparation, of de novo or restenotic lesions up to 180 mm in length in native superficial femoral or popliteal arteries with reference vessel diameters of 4-6 mm.
  Interventions: Device: Stellarex 0.035" OTW Drug-coated Angioplasty Balloon
- PTA Subjects (Placebo Comparator): The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA).
  Basic Catheter Specifications
  * Guidewire: 0.035"
  * Balloon Length: 40/80/120 mm
  * Sheath Compatibility: greater to or equal to 6 French
  * Balloon Diameter: 4/5/6 mm
  * Shaft length: 135 cm Indications The EverCross Balloon Catheter is intended to dilate stenosis in the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries, and to treat obstructive lesions of native or synthetic arteriovenous dialysis fistulae. This device is also indicated for stent post-dilation in the peripheral vasculature. For additional information refer to the EverCross Instructions for Use.
  Interventions: Device: EverCross™ 0.035 PTA Balloon Catheter

INTERVENTIONS:
Device: Stellarex 0.035" OTW Drug-coated Angioplasty Balloon — The Stellarex 0.035" OTW Drug-coated Angioplasty Balloon is indicated for percutaneous transluminal angioplasty (PTA), after appropriate vessel preparation, of de novo or restenotic lesions up to 180 mm in length in native superficial femoral or popliteal arteries with reference vessel diameters of 4-6 mm.
  Arms: DCB Subjects
Device: EverCross™ 0.035 PTA Balloon Catheter — The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA).
  Arms: PTA Subjects

SUMMARY:
The ILLUMENATE Pivotal PAS is a continued follow-up study which will include 300 subjects from forty-three (43) sites across the United States and Austria previously enrolled in the ILLUMENATE Pivotal pre-market study to evaluate the Stellarex DCB compared to the PTA control device for the treatment of de-novo or post-PTA occluded/stenotic or reoccluded/restenotic (except for in-stent) SFA and/or popliteal arteries.

DETAILED DESCRIPTION:
The objective of this continued follow-up of ILLUMENATE Pivotal Study subjects is to demonstrate the long term safety and effectiveness of the Stellarex DCB.

Each enrolled subject will be followed for 5 years (60 months) after treatment. A follow-up office visit will occur at 24 and 36 months. A follow-up telephone contact or an optional office visit will occur at 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria - From ILLUMENATE Pivotal IDE population TP-1397E

Study subjects must fulfill the following clinical criteria:

1. Symptomatic leg ischemia, requiring treatment of the superficial femoral artery (SFA) and/or popliteal artery.
2. Greater than or equal to 18 years of age.
3. Willing to provide written informed consent, and capable and willing to comply with all required follow-up evaluations within the defined follow-up visit windows.
4. Will not undergo other planned vascular interventions within 14 days before and/or 30 days after the protocol treatment (successful treatment of ipsilateral and contralateral iliac permitted prior to enrollment).
5. Life expectancy >1 year.
6. Rutherford-Becker classification of 2, 3 or 4.

   Study Subjects must fulfill the following angiographic criteria:
7. De novo or restenotic lesion (except for in-stent restenotic lesion) >70% within the SFA and/or popliteal artery in a single limb.
8. Single lesion which is ≥3 cm and ≤18cm in length (by visual estimation). NOTE: Tandem lesions can be treated. A tandem lesion is defined as two distinct lesions with 3 cm or less of healthy vessel separating the two diseased areas. The total cumulative length of the tandem lesions, including the healthy vessel, must not exceed 18 cm.
9. Lesion is treatable by no more than two (2) study devices.
10. Successful wire crossing of the lesion. The guidewire advancement should not be indicative of the presence of fresh thrombus in the lesion.
11. Target reference vessel diameter is ≥4 mm and ≤6 mm (by visual estimation).
12. Inflow artery is patent, free from significant lesion stenosis (≥50% stenosis is considered significant) as confirmed by angiography. Treatment of a target lesion is acceptable after successful treatment of inflow artery lesion(s). NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis <30% without death or major vascular complication.
13. Target limb with at least one patent (less than 50% stenosis) tibio-peroneal run-off vessel confirmed by baseline angiography or prior magnetic resonance (MR) angiography or computed tomography (CT) angiography (within 45 days prior to index procedure). NOTE: treatment of outflow disease is NOT permitted.

Exclusion Criteria -

Subject with any of the following clinical criteria should be excluded:

1. Females who are pregnant, lactating, or intend to become pregnant, or males who intend to father children during study participation.
2. Known aortic aneurysm(s) > 5 cm.
3. Contraindication to dual anti-platelet therapy.
4. Known intolerance to study medications, paclitaxel or contrast agents that in the opinion of the investigator cannot be adequately pre-treated.
5. Current participation in an investigational drug or another device study.
6. History of hemorrhagic stroke within 3 months.
7. Previous or planned surgical or interventional procedure within 14 days before or 30 days after the index procedure (successful treatment of ipsilateral and contralateral iliac permitted prior to enrollment).
8. Prior endovascular treatment of target lesion by percutaneous transluminal angioplasty or any other means of previous endovascular treatment (e.g. stents/stent grafts, cutting balloon, scoring balloon, cryoplasty, thrombectomy, atherectomy, brachytherapy or laser devices) within six months of the index procedure, or any previous placement of a bypass graft proximal to the target lesion.
9. Treatment of lesions in the contralateral limb with the CVI Paclitaxel-coated PTA Catheter.
10. Use of the CVI Paclitaxel-coated PTA Catheter in other than a single treatment session.
11. Chronic renal insufficiency (dialysis dependent, or serum creatinine >2.5 mg/dL within 30 days of index procedure).

    Subject with any of the following angiographic criteria should be excluded:
12. Significant contralateral or ipsilateral common femoral disease that requires intervention during the index procedure.
13. No normal proximal arterial segment of the target vessel in which duplex ultrasound velocity ratios can be measured.
14. Known inadequate distal outflow.
15. Acute or sub-acute thrombus in the target vessel.
16. Aneurysmal target vessel.
17. Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloons, brachytherapy) during the index procedure in the target lesion or target vessel.
18. Treatment of the contralateral limb during the same procedure or within 30 days following the study procedure (exclusive of the iliac arteries which can be treated prior to enrollment).
19. Presence of concentric calcification that precludes PTA pre-dilation.
20. Prior stent placement in the target vessel.
21. Residual stenosis of greater than 70%, stent placement or flow-limiting (Grade D or greater) dissection following pre-dilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lyden, MD, Principal Investigator — The Cleveland Clinic; Prakash Krishnan, MD, Principal Investigator — Mount Sinai Health System
Locations (41):
- United States (39):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Mission Cardiovascular Research Institute, Fremont, California
  - Good Samaritan Hospital - Los Angeles, Los Angeles, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Cardiovascular Research of North Florida, Gainesville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Central Iowa Hospital Corporation, Des Moines, Iowa
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Wake Heart Research, Raleigh, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - North Ohio Research LTD., Elyria, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Heritage Valley Health System, Beaver, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, INC., Wormleysburg, Pennsylvania
  - Sanford Health Vascular Associates, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Wellmont Holston Valley Medical, Kingsport, Tennessee
  - Premier Surgical Associates, Knoxville, Tennessee
  - Texas Health & Research Education Institution, Dallas, Texas
  - El Paso Cardiology Associates, El Paso, Texas
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - CAMC Clinical Trial Center, Charleston, West Virginia
  - Aurora Health Care, Milwaukee, Wisconsin
- Austria (2):
  - Medical University Graz, Graz
  - Hanusch Krankenhaus Wien, Vienna

REFERENCES:
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024

RESULTS

PARTICIPANT FLOW:
Groups:
- DCB Subjects: The Stellarex DCB is a commercially available PTA balloon catheter (EverCross™ 0.035" PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA) coated with paclitaxel using a proprietary carrier.
  Basic Catheter Specifications
  * Guidewire: 0.035"
  * Balloon Length: 40/80/120 mm
  * Sheath Compatibility: greater than or equal to 6 French
  * Balloon Diameter: 4/5/6 mm
  * Shaft length: 135 cm The nominal dose density of paclitaxel on the Stellarex DCB is 2.0 μg/mm2. Indications The Stellarex 0.035" OTW Drug-coated Angioplasty Balloon is indicated for percutaneous transluminal angioplasty (PTA), after appropriate vessel preparation, of de novo or restenotic lesions up to 180 mm in length in native superficial femoral or popliteal arteries with reference vessel diameters of 4-6 mm.
  Stellarex 0.035" OTW Drug-coated Angioplasty Balloon: The Stellarex 0.035" OTW Drug-coated Angioplasty Balloon is indicated for percutaneous transluminal angioplasty (PTA), after appropriate vessel preparation, of de novo or restenotic lesions up to 180 mm in length in native superficial femoral or popliteal arteries with reference vessel diameters of 4-6 mm.
- PTA Subjects: The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA).
  Basic Catheter Specifications
  * Guidewire: 0.035"
  * Balloon Length: 40/80/120 mm
  * Sheath Compatibility: greater to or equal to 6 French
  * Balloon Diameter: 4/5/6 mm
  * Shaft length: 135 cm Indications The EverCross Balloon Catheter is intended to dilate stenosis in the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries, and to treat obstructive lesions of native or synthetic arteriovenous dialysis fistulae. This device is also indicated for stent post-dilation in the peripheral vasculature. For additional information refer to the EverCross Instructions for Use.
  EverCross™ 0.035 PTA Balloon Catheter: The control device is a commercially available PTA balloon catheter (EverCross™ 0.035 PTA Balloon Catheter, Medtronic, Plymouth, MN 55441, USA).
Period: Overall Study
Arm/Group | DCB Subjects | PTA Subjects
Started | 200 | 100
Completed | 135 | 70
Not Completed | 65 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCB Subjects | PTA Subjects | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.3) | 69.8 (9.8) | 68.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 36 | 124
  Male | 112 | 64 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all participants reported this demographic information.
  Participants
    Hispanic or Latino | 27 | 11 | 38
    Not Hispanic or Latino | 152 | 77 | 229
    Unknown or Not Reported | 21 | 12 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all participants reported this demographic.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | NA — Native Hawaiian or Pacific Islander was not collected. | NA — Native Hawaiian or Pacific Islander was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Black or African American | 35 | 19 | 54
    White | 142 | 68 | 210
    More than one race | NA — More than one race was not collected. | NA — More than one race was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Unknown or Not Reported | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  Austria | 17 | 10 | 27
  United States | 183 | 90 | 273
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (6.1) | 28.8 (5.6) | 29.0 (6.0)
Ankle-Brachial Index [Mean (Standard Deviation); unit: ratio] — Population: Data was analyzed by arm, not by total. ABI analysis returns measurement values of mmHg. Non-compressible indicates no measurement could be taken, therefore there is no measurement to analyze and report.
  ratio
    Ankle-Brachial Index Measurement: number analyzed (Participants) | 193 | 100 | 293
    Ankle-Brachial Index Measurement | 0.75 (0.21) | 0.76 (0.20) | 0.75 (0.21)
    Non-Compressible: number analyzed (Participants) | 6 | 0 | 6
    Non-Compressible | NA (NA) — Non-compressible does not return a measurement, no value is available. |  | NA (NA) — Non-compressible does not return a measurement, no value is available.
Rutherford-Becker Clinical Category [Count of Participants; unit: Participants]
  RCC 2 | 63 | 35 | 98
  RCC 3 | 129 | 60 | 189
  RCC 4 | 8 | 5 | 13
Peripheral Vascular Disease (PVD) [Count of Participants; unit: Participants] | 200 | 100 | 300
Hypertension [Count of Participants; unit: Participants] | 187 | 94 | 281
Hyperlipidemia [Count of Participants; unit: Participants] | 176 | 90 | 266
Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 42 | 22 | 64
Angina Pectoris [Count of Participants; unit: Participants] | 30 | 20 | 50
Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 24 | 8 | 32
Previous Percutaneous or Surgical Coronary Revascularization [Count of Participants; unit: Participants] | 90 | 48 | 138
Renal Insufficiency [Count of Participants; unit: Participants] | 36 | 17 | 53
Liver Disease [Count of Participants; unit: Participants] | 7 | 4 | 11
Cerebrovascular Disease [Count of Participants; unit: Participants] | 47 | 20 | 67
Chronic Obstructive Pulmonary Occlusion (COPD) [Count of Participants; unit: Participants] | 32 | 21 | 53
Deep Vein Thrombosis (DVT) [Count of Participants; unit: Participants] | 6 | 4 | 10
Diabetes (Total) [Count of Participants; unit: Participants] | 99 | 52 | 151
Diabetes - Type I [Count of Participants; unit: Participants] | 8 | 3 | 11
Diabetes - Type II [Count of Participants; unit: Participants] | 91 | 49 | 140
Smoker [Count of Participants; unit: Participants]
  Never Smoked | 32 | 24 | 56
  Previous or Current Smoker | 168 | 76 | 244
Previous Intervention of the Lower Limb [Count of Participants; unit: Participants] | 87 | 41 | 128
Previous Intervention of the Study Limb [Count of Participants; unit: Participants] | 48 | 23 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Patency at 24 Months Post-procedure
Description: Patency is defined as the absence of target lesion restenosis as determined by duplex ultrasound (Peak Systolic Velocity Ratio (PSVR) ≤ 2.5) and freedom from clinically-driven target lesion revascularization.
Time Frame: 24 months post-procedure
Population: Patency was defined as absence of target lesion restenosis (as assessed by the duplex ultrasound core laboratory based on PSVR ≤ 2.5) and CD-TLR through 24 months (defined as 730 ± 45 days, i.e., up to 775 days) or angiographic core laboratory assessment of restenosis. Denominators represent the number of intent-to-treat participants from each arm for whom data are available for this outcome (200 DCB and 100 PTA were enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 146 | 87
Participants | 88 | 45

2. Primary Outcome: Number of Participants With Freedom From Device and Procedure Related Death Through 30 Days Post-procedure and Freedom From Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization Through 24 Months Post-procedure
Description: The primary safety outcome is defined as freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation and clinically-driven target lesion revascularization (CD-TLR) through 24 months post-procedure (defined as 730 ± 45 days, i.e., up to 775 days).
Time Frame: 24 months post-procedure
Population: Subject was considered a failure if they experienced device or procedure-related death within 30 days, or if they experienced target limb major amputation or CD-TLR within 24 months (defined as 730 ± 45 days, i.e., up to 775 days). Denominators represent the number of intent-to-treat participants from each arm for whom data are available for this outcome (200 DCB and 100 PTA were enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 171 | 92
Participants | 142 | 73

3. Secondary Outcome: Major Adverse Event (MAE) Rate at 24 Months Post-procedure, Defined as a Composite Rate of Cardiovascular Death, Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization (TLR)
Description: Major adverse event (MAE) rate at 24 months post-procedure, defined as a composite rate of cardiovascular death, target limb major amputation and clinically-driven target lesion revascularization (TLR).
Time Frame: 24 months post-procedure
Population: Denominators represent the number of intent-to-treat participants from each arm for whom data are available for this outcome (200 DCB and 100 PTA were enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 183 | 94
Participants | 34 | 22

4. Secondary Outcome: Major Adverse Event (MAE) Rate at 36 Months Post-procedure, Defined as a Composite Rate of Cardiovascular Death, Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization (TLR)
Description: Major adverse event (MAE) rate at 36 months post-procedure, defined as a composite rate of cardiovascular death, target limb major amputation and clinically-driven target lesion revascularization (TLR).
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 176 | 91
Participants | 46 | 27

5. Secondary Outcome: Major Adverse Event (MAE) Rate at 48 Months Post-procedure, Defined as a Composite Rate of Cardiovascular Death, Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization (TLR)
Description: Major adverse event (MAE) rate at 48 months post-procedure, defined as a composite rate of cardiovascular death, target limb major amputation and clinically-driven target lesion revascularization (TLR).
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 166 | 88
Participants | 55 | 33

6. Secondary Outcome: Major Adverse Event (MAE) Rate at 60 Months Post-procedure, Defined as a Composite Rate of Cardiovascular Death, Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization (TLR)
Description: Major adverse event (MAE) rate at 60 months post-procedure, defined as a composite rate of cardiovascular death, target limb major amputation and clinically-driven target lesion revascularization (TLR).
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 156 | 83
Participants | 64 | 37

7. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization
Description: Lesion revascularization occuring in the target lesion deemed clinically driven by the Clinical Events Committee. Clinically-driven target lesion revascularization is a repeat revascularization procedure at the target lesion due to a peak systolic velocity ratio ≥ 2.5 by duplex ultrasound or a percent diameter stenosis >50% by angiography accompanied by worsening of the Rutherford Becker Clinical Category or Ankle Brachial Index that is clearly referable to the target lesion.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 179 | 92
Participants | 29 | 19

8. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization
Description: Lesion revascularization occurring in the target lesion deemed clinically driven by the Clinical Events Committee. Clinically-driven target lesion revascularization is a repeat revascularization procedure at the target lesion due to a peak systolic velocity ratio ≥ 2.5 by duplex ultrasound or a percent diameter stenosis >50% by angiography accompanied by worsening of the Rutherford Becker Clinical Category or Ankle Brachial Index that is clearly referable to the target lesion.
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 170 | 88
Participants | 38 | 24

9. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization
Description: as for outcome 7
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 158 | 83
Participants | 44 | 28

10. Secondary Outcome: Rate of Clinically-driven Target Lesion Revascularization
Description: as for outcome 8
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 143 | 75
Participants | 51 | 29

11. Secondary Outcome: Rate of Target Lesion Revascularization
Description: Lesion revascularization occuring in the target lesion deemed clinically driven by the Clinical Events Committee
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 180 | 92
Participants | 32 | 20

12. Secondary Outcome: Rate of Target Lesion Revascularization
Description: Lesion revascularization occuring in the target lesion deemed clinically driven by the Clinical Events Committee
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 171 | 88
Participants | 42 | 25

13. Secondary Outcome: Rate of Target Lesion Revascularization
Description: Lesion revascularization occuring in the target lesion deemed clinically driven by the Clinical Events Committee
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 159 | 83
Participants | 48 | 29

14. Secondary Outcome: Rate of Target Lesion Revascularization
Description: Lesion revascularization occuring in the target lesion deemed clinically driven by the Clinical Events Committee
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 144 | 76
Participants | 55 | 30

15. Secondary Outcome: Rate of Clinically-driven Target Vessel Revascularization
Description: Lesion revascularization occuring in the target vessel deemed clinically driven by the Clinical Events Committee. A clinically-driven target vessel revascularization is a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. A revascularization of the target vessel is considered clinically-driven if the peak systolic velocity ratio ≥ 2.5 by duplex ultrasound or if angiography shows a percent diameter stenosis >50% and there is worsening of the Rutherford Becker Clinical Category or Ankle-Brachial Index.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 178 | 91
Participants | 1 | 1

16. Secondary Outcome: Rate of Clinically-driven Target Vessel Revascularization
Description: Lesion revascularization occurring in the target vessel deemed clinically driven by the Clinical Events Committee. A clinically-driven target vessel revascularization is a repeat revascularization procedure (percutaneous or surgical) of a lesion in the target vessel, exclusive of the target lesion site. A revascularization of the target vessel is considered clinically-driven if the peak systolic velocity ratio ≥ 2.5 by duplex ultrasound or if angiography shows a percent diameter stenosis >50% and there is worsening of the Rutherford Becker Clinical Category or Ankle-Brachial Index.
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 169 | 83
Participants | 3 | 1

17. Secondary Outcome: Rate of Clinically-driven Target Vessel Revascularization
Description: as for outcome 16
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 155 | 78
Participants | 3 | 2

18. Secondary Outcome: Rate of Clinically-driven Target Vessel Revascularization
Description: as for outcome 16
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 135 | 67
Participants | 3 | 2

19. Secondary Outcome: Rate of Target Limb Major Amputation
Description: Number of subjects in which a major amputation occurred in the target limb
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 178 | 91
Participants | 1 | 0

20. Secondary Outcome: Rate of Target Limb Major Amputation
Description: Number of subjects in which a major amputation occurred in the target limb
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 169 | 83
Participants | 1 | 0

21. Secondary Outcome: Rate of Target Limb Major Amputation
Description: Number of subjects in which a major amputation occurred in the target limb
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 155 | 78
Participants | 2 | 0

22. Secondary Outcome: Rate of Target Limb Major Amputation
Description: Number of subjects in which a major amputation occurred in the target limb
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 137 | 67
Participants | 2 | 0

23. Secondary Outcome: Mortality Rate
Description: Number of subject who have died during the post-procedure follow up period
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 190 | 97
Participants | 13 | 8

24. Secondary Outcome: Mortality Rate
Description: Number of subject who have died during the post-procedure follow up period
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 185 | 93
Participants | 18 | 10

25. Secondary Outcome: Mortality Rate
Description: Number of subject who have died during the post-procedure follow up period
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 178 | 91
Participants | 27 | 14

26. Secondary Outcome: Mortality Rate
Description: Number of subject who have died during the post-procedure follow up period
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 169 | 86
Participants | 34 | 19

27. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Description: Rate of occurrence of arterial thrombosis of the treated segment
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 178 | 91
Participants | 3 | 0

28. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Description: Rate of occurrence of arterial thrombosis of the treated segment
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 169 | 83
Participants | 4 | 0

29. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Description: Rate of occurrence of arterial thrombosis of the treated segment
Time Frame: 48 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 155 | 78
Participants | 4 | 0

30. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Description: Rate of occurrence of arterial thrombosis of the treated segment
Time Frame: 60 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 135 | 67
Participants | 4 | 0

31. Secondary Outcome: Patency Rate Defined as the Absence of Target Lesion Restenosis as Determined by Duplex Ultrasound (PSVR ≤ 2.5) and Freedom From Clinically-driven TLR
Description: Patency rate defined as the absence of target lesion restenosis as determined by duplex ultrasound (PSVR ≤ 2.5) and freedom from clinically-driven TLR
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 146 | 87
Participants | 88 | 45

32. Secondary Outcome: Patency Rate Defined as the Absence of Target Lesion Restenosis as Determined by Duplex Ultrasound (PSVR ≤ 2.5) and Freedom From Clinically-driven TLR
Description: as for outcome 31
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 116 | 73
Participants | 65 | 35

33. Secondary Outcome: Change in Ankle-brachial Index (ABI) From Pre-procedure
Description: The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). The normal range for the ankle-brachial index is between 0.90 and 1.30. An index under 0.90 means that blood is having a hard time getting to the legs and feet: 0.41 to 0.90 indicates mild to moderate peripheral artery disease; 0.40 and lower indicates severe disease.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 141 | 79
Participants
  Improved | 102 | 56
  No Change | 0 | 1
  Worsened | 39 | 22

34. Secondary Outcome: Change in Ankle-brachial Index (ABI) From Pre-procedure
Description: as for outcome 33
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 120 | 69
Participants
  Improved | 89 | 46
  Worsened | 31 | 23

35. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) From Pre-procedure
Description: A disease-specific instrument utilized to characterize walking ability through a questionnaire. It is a measure of patient-perceived walking performance for patients with PAD and/or intermittent claudication
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 153 | 82
Participants
  Improved | 114 | 63
  Worsened | 39 | 19

36. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) From Pre-procedure
Description: as for outcome 35
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 131 | 74
Participants
  Improved | 98 | 50
  No Change | 1 | 0
  Worsened | 32 | 24

37. Secondary Outcome: Change in Walking Distance From Pre-procedure
Description: Distance in meters or feet traveled in 6 minutes measured at pre-procedure and at 24 month office visit.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 142 | 80
Participants
  Improved | 92 | 57
  No Change | 1 | 1
  Worsened | 49 | 22

38. Secondary Outcome: Change in Walking Distance From Pre-procedure
Description: Distance in meters or feet traveled in 6 minutes measured at pre-procedure and at 36 month office visit.
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 114 | 69
Participants
  Improved | 77 | 47
  No Change | 2 | 0
  Worsened | 35 | 22

39. Secondary Outcome: Change in Rutherford-Becker Classification From Pre-procedure
Description: Rutherford-Becker Classification is a classification system of Peripheral Arterial Disease, the higher the number the worse the disease.
  Category Clinical Description 0-Asymptomatic--no hemodynamically significant occlusive disease
  Mild claudication Moderate claudication Severe claudication 4*-Ischemic rest pain 5*-Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia 6*-Major tissue loss-extending above transmetatarsal level, functional foot no longer salvageable *Categories 4, 5, and 6 are also described as critical limb ischemia.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 153 | 82
Participants
  Improved | 128 | 74
  No Change | 17 | 5
  Worsened | 8 | 3

40. Secondary Outcome: Change in Rutherford-Becker Classification From Pre-procedure
Description: as for outcome 39
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 130 | 76
Participants
  Improved | 108 | 63
  No Change | 15 | 11
  Worsened | 7 | 2

41. Secondary Outcome: Change in EQ-5D Index From Pre-procedure
Description: EQ-5D is designed for self-completion by subjects and is intended to reflect the health status at the time of completion.
Time Frame: 24 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 103 | 59
Participants
  Improved | 62 | 37
  No Change | 9 | 7
  Worsened | 32 | 15

42. Secondary Outcome: Change in EQ-5D Index From Pre-procedure
Description: as for outcome 41
Time Frame: 36 months post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 95 | 56
Participants
  Improved | 52 | 35
  No Change | 15 | 6
  Worsened | 28 | 15

43. Secondary Outcome: Change in EQ-5D VAS From Pre-procedure
Description: as for outcome 41
Time Frame: 24 months post procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 104 | 59
Participants
  Improved | 52 | 30
  No Change | 12 | 10
  Worsened | 40 | 19

44. Secondary Outcome: Change in EQ-5D VAS From Pre-procedure
Description: as for outcome 41
Time Frame: 36 month post procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | DCB Subjects | PTA Subjects
Number analyzed (Participants) | 95 | 56
Participants
  Improved | 53 | 26
  No Change | 6 | 9
  Worsened | 36 | 21

ADVERSE EVENTS:
Time Frame: Adverse Event reporting begins at the time the subject is enrolled in the study and continues through their exit which can be as long as 60 months. Please note these patients are a roll-over from NCT01858428 and continues the subjects follow-up.
Description: The definitions are the same.
Arm/Group | DCB Subjects | PTA Subjects
All-Cause Mortality (participants affected / at risk) | 34/200 | 19/100
Serious Adverse Events (participants affected / at risk) | 177/200 | 85/100
Other Adverse Events (participants affected / at risk) | 192/200 | 95/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCB Subjects (N=200) | PTA Subjects (N=100)
Anaemia (Blood and lymphatic system disorders) | 8 (12) | 3 (3)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypchromic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 7 (11) | 3 (3)
Angina Pectoris (Cardiac disorders) | 11 (14) | 2 (3)
Angina Unstable (Cardiac disorders) | 5 (7) | 2 (2)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 8 (10) | 6 (13)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 2 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 6 (6) | 1 (10)
Cardiac Failure Acute (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 12 (20) | 5 (6)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 12 (14) | 4 (5)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 4 (4) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetance (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Torsade de Pointes (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (3)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blindness Unilateral (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Macular Fibrosis (Eye disorders) | 1 (1) | 0 (0)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 3 (3)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Angiodysplasia Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 7 (7) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 4 (5) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small Intestine Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter Site Hematoma (General disorders) | 1 (1) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 20 (30) | 8 (8)
Death (General disorders) | 4 (4) | 6 (6)
Device Deployment Issue (General disorders) | 1 (1) | 0 (0)
Device Occlusion (General disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1)
Medical Device Complication (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 4 (5) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Vessel Puncture Site Thrombosis (General disorders) | 1 (1) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelthiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis Perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (3) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bursitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 5 (9) | 3 (4)
Device Related Infection (Infections and infestations) | 2 (2) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Enfocarditis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 2 (3) | 0 (0)
FUNGAEMIA (Infections and infestations) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GROIN ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
H1N1 INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CORONARY BYPASS THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GRAFT HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 24 (33) | 13 (19)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 2 (3) | 0 (0)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (12) | 3 (3)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CERVIX CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
SPLENIC NEOPLASM MALIGNANCY UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 6 (10) | 4 (5)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2 (2) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 5 (6) | 1 (1)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
CERVICAL MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 3 (5)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 4 (4)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
IVTH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
POSTICTAL STATE (Nervous system disorders) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 7 (7) | 5 (5)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 (4) | 1 (1)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 (0) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (2) | 0 (0)
DEPENDENCE (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (2) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (2) | 2 (2)
INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2 (2) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 3 (3) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 14 (17) | 3 (5)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 4 (5) | 1 (2)
URINARY RETENTION (Renal and urinary disorders) | 3 (3) | 0 (0)
URINARY TRACT INFLAMMATION (Renal and urinary disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infected Seroma (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pasteurella Infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 14 (20) | 9 (10)
Sepsis (Infections and infestations) | 5 (6) | 4 (4)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 7 (9) | 3 (3)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANGIOPLASTY (Surgical and medical procedures) | 2 (2) | 0 (0)
AORTIC VALVE REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1)
CATARACT OPERATION (Surgical and medical procedures) | 1 (2) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 2 (3) | 0 (0)
OBESITY SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
PERIPHERAL ARTERY BYPASS (Surgical and medical procedures) | 0 (0) | 1 (1)
PERIPHERAL REVASCULARISATION (Surgical and medical procedures) | 1 (1) | 2 (2)
RESECTION OF RECTUM (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
TOE AMPUTATION (Surgical and medical procedures) | 2 (2) | 0 (0)
WOUND DRAINAGE (Surgical and medical procedures) | 1 (1) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 3 (3) | 2 (2)
AORTIC STENOSIS (Vascular disorders) | 6 (6) | 0 (0)
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL STENOSIS (Vascular disorders) | 1 (1) | 1 (1)
BLUE TOE SYNDROME (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 17 (17) | 6 (6)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 5 (6) | 2 (3)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 5 (5) | 2 (2)
HYPERTENSIVE CRISIS (Vascular disorders) | 3 (3) | 2 (2)
HYPOTENSION (Vascular disorders) | 6 (7) | 2 (2)
INTERMITTENT CLAUDICATION (Vascular disorders) | 43 (59) | 18 (23)
ISCHAEMIA (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 9 (10) | 2 (2)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 45 (64) | 27 (42)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 4 (4) | 0 (0)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 6 (6) | 1 (1)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 1 (1)
VENOUS INSUFFICIENCY (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCB Subjects (N=200) | PTA Subjects (N=100)
Anaemia (Blood and lymphatic system disorders) | 16 (21) | 6 (7)
Angina Pectoris (Cardiac disorders) | 14 (19) | 6 (7)
Atrial Fibrillation (Cardiac disorders) | 12 (16) | 11 (20)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 13 (21) | 6 (8)
CORONARY ARTERY DISEASE (Cardiac disorders) | 14 (16) | 5 (6)
CATARACT (Eye disorders) | 2 (3) | 5 (7)
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 (15) | 6 (6)
CHEST PAIN (General disorders) | 35 (55) | 17 (23)
LOCAL SWELLING (General disorders) | 7 (8) | 10 (13)
OEDEMA PERIPHERAL (General disorders) | 13 (13) | 11 (13)
BRONCHITIS (Infections and infestations) | 12 (13) | 3 (3)
CELLULITIS (Infections and infestations) | 9 (13) | 6 (8)
PNEUMONIA (Infections and infestations) | 18 (24) | 10 (11)
URINARY TRACT INFECTION (Infections and infestations) | 20 (25) | 7 (11)
CONTUSION (Injury, poisoning and procedural complications) | 17 (23) | 3 (4)
FALL (Injury, poisoning and procedural complications) | 5 (8) | 5 (5)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 30 (41) | 18 (25)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 20 (27) | 15 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 20 (23) | 9 (11)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 16 (18) | 7 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (10) | 7 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 48 (64) | 21 (23)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 7 (13) | 6 (7)
DIZZINESS (Nervous system disorders) | 10 (12) | 3 (7)
HEADACHE (Nervous system disorders) | 10 (15) | 2 (4)
SYNCOPE (Nervous system disorders) | 10 (12) | 7 (7)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 19 (22) | 5 (8)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 11 (29) | 6 (10)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 29 (37) | 11 (19)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (6)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (6)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 17 (19) | 6 (6)
HAEMATOMA (Vascular disorders) | 13 (14) | 3 (3)
HYPERTENSION (Vascular disorders) | 12 (14) | 6 (9)
HYPOTENSION (Vascular disorders) | 10 (14) | 2 (5)
INTERMITTENT CLAUDICATION (Vascular disorders) | 74 (124) | 35 (56)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 13 (16) | 6 (7)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 54 (98) | 34 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Institution and PI shall have the right to publish, present or otherwise publicly disclose the results to their own activity conducted in the trial. Proposals must be submitted to the sponsor for review 30 days prior to publishing submission. Sponsor has the right to require confidentially sensitive information be removed (not including results) and/or delay publication for an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03421561/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03421561/SAP_002.pdf